CLINICAL TRIAL: NCT07286565
Title: Active-NBS Liege - Monitoring the Motor Development of Children With Duchenne Muscular Dystrophy or Spinal Muscular Atrophy Identified Through Newborn Screening
Brief Title: Active NBS Study: Decentralised Monitoring Motor Development in Children With Duchenne Muscular Dystrophy or Spinal Muscular Atrophy Identified by Newborn Screening
Acronym: Active-NBS BE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry); Centre Hospitalier Régional de la Citadelle (Other); Leon Fredericq Foundation (Unknown)
Responsible Party: Principal Investigator, Tamara DANGOULOFF, Dr, Centre Hospitalier Universitaire de Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Active-NBS Liege
Record Dates: First submitted 2025-09-05; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy (SMA); Duchenne Muscular Dystrophy (DMD)
Keywords: Remotely monitor; Syde; Accelerometry; Daily living
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Dystrophy, Duchenne | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with spinal muscular atrophy (Experimental): Patients will wear a device (Maiju and/or Syde) and complete questionnaires.
  Interventions: Device: MAIJU; Device: Syde; Other: Questionnaires; Other: PedsQL Questionnaire
- Patient with Duchenne muscular disease (Experimental): Patients will wear a device (Maiju and/or Syde) and complete questionnaires.
  Interventions: Device: MAIJU; Device: Syde; Other: Questionnaires; Other: PedsQL Questionnaire

INTERVENTIONS:
Device: MAIJU — A jumpsuit equipped with motion sensors for detailed assessment of motor development and postural changes. Developed by the University of Helsinki, it enables remote evaluation of infants and their motor behavior. The device has been extensively validated in healthy infants and those with cerebral palsy
Device: Syde — The Syde® is a Class I medical device, CE-marked (compliant with European Regulation 2017/745) and manufactured by Sysnav (Vernon, France). The Syde® measures various gait parameters to assess motor abilities. It enabled the identification of SV95C in Duchenne muscular dystrophy (DMD), which became the first qualified primary endpoint in DMD, and the first digital outcome qualified by a regulatory agency. Data have been collected in about thirty DMD children under 4 years old and in an age-matched control population. These data demonstrated feasibility, reliability, and sensitivity to change in children from controls as soon as walking is acquired.
Other: Questionnaires — Parents will complete a specific questionnaire covering their child's medical history;
Other: PedsQL Questionnaire — Quality-of-life questionnaire

SUMMARY:
The Active NBS Liege study is a monocentric, academic, fully remote, observational study designed to validate digital measures of motor development in children with spinal muscular atrophy (SMA) or Duchenne muscular dystrophy (DMD) identified through newborn screening, family testing, or incidental diagnosis. The study will enroll 100 children and follow them longitudinally for up to 30 months. Participants are remotely recruited, and all procedures, including consent, questionnaires, and follow-up visits, are conducted by phone or video conferencing without any hospital visits. Children will use age-appropriate wearable devices at home: MAIJU®, a sensorized garment for non-ambulant infants, and Syde®, an ankle-worn sensor for ambulant children. Data collection includes digital motor endpoints, clinical information, and quality of life (PedsQL). Primary objectives are to validate digital biomarkers of motor development, while secondary objectives include early identification of motor deficits, modeling motor trajectories, and quantifying genotype-related differences. Exploratory analyses will assess gait parameters such as stride velocity 95th centile (SV95C) and compare motor outcomes across genetic profiles and treatment exposure. Risks are minimal, limited to the use of non-invasive sensors with no known side effects.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) and spinal muscular atrophy (SMA) are severe, progressive, and life-limiting neuromuscular disorders that manifest during early childhood. Both conditions are characterized by motor function decline, leading to severe disability and premature mortality. The availability of disease-modifying therapies has dramatically changed the clinical landscape, but their effectiveness is strongly dependent on very early initiation, ideally before symptom onset.

Newborn screening (NBS) for SMA has now been implemented in several countries, enabling the identification of affected infants at birth. This shift creates a new challenge: the need to monitor presymptomatic or minimally symptomatic children over time with sensitive, reliable, and age-appropriate tools. Conventional motor function scales were designed for older children and are not sufficiently adapted for infants and toddlers. As a result, there is a critical gap in longitudinal assessment during the first years of life, a period when therapeutic interventions may have the greatest impact.

The Active NBS study was designed to address this unmet need. This is a monocentric, fully remote, academic, observational study that leverages wearable digital technologies to monitor motor development in very young children with SMA or DMD. The study is conducted entirely at a distance, with no requirement for hospital visits, thereby reducing the burden on families and improving accessibility.

Study Objectives:

The primary objective is to validate digital biomarkers of early motor development in children diagnosed with SMA or DMD. Secondary objectives include the early detection of motor deficits, quantification of developmental delays according to genetic subtype, and modeling of motor trajectories during the first years of life. Exploratory objectives focus on gait analysis, including stride velocity 95th centile (SV95C), and comparisons of motor outcomes across genetic backgrounds and treatment exposure.

Study Design and Procedures:

Up to 100 children will be enrolled, including infants identified by NBS, family testing, or incidental diagnosis. Enrollment and informed consent are performed remotely using secure electronic platforms. Participants are followed prospectively for up to 30 months, with assessments every 6 months through structured questionnaires and video consultations with the study team.

Two wearable devices will be employed, depending on the child's age and motor status:

* MAIJU® (Motor Assessment of Infants with a Jumpsuit): a sensorized garment designed for non-ambulant infants, capturing spontaneous movement and generating a composite biomarker (Babacloud Infant Motility Score, BIMS).
* Syde®: a wearable ankle sensor validated in ambulant children, enabling precise gait monitoring and calculation of SV95C, a regulatory-accepted endpoint in DMD.

Data collected include digital motor endpoints, routine clinical information, and quality of life metrics (PedsQL). Families are instructed on the correct use of devices and can install and remove them independently at home. No travel or in-person assessments are required, making this approach particularly suitable for rare disease populations.

Scientific Rationale:

Traditional motor scales, while validated in older children, lack sensitivity to detect subtle developmental changes in infancy and early childhood. Digital endpoints derived from continuous movement monitoring have the potential to provide richer, objective data on motor development. By validating these measures in a presymptomatic or early symptomatic population, this study aims to establish novel tools for both clinical practice and future interventional trials. Importantly, the study also addresses the practical and ethical challenges of long-term follow-up in very young children by implementing a fully remote design.

Expected Impact:

The Active NBS study is expected to generate the first large-scale, longitudinal dataset on motor development in presymptomatic and early symptomatic children with SMA and DMD. The validation of digital endpoints such as SV95C and BIMS will contribute to the development of sensitive outcome measures for clinical trials and may support regulatory acceptance in the future. Beyond its immediate scientific goals, the study demonstrates the feasibility and acceptability of decentralized follow-up in rare pediatric populations, setting the stage for broader applications of digital health technologies in neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

Genetically confirmed SMA and avalaible MSNA2 copy number:

* Identified by newborn screening,
* Identified by family screening, or incidental diagnosis in pre-symptomatic stage
* Treated (or follow-up possible for patients with 4 SMN2 copies)

Genetically confirmed DMD:

* Identified by newborn screening,
* Identified by family screening, or incidental diagnosis in pre-symptomatic stage
* Age < 4 years at inclusion

Legal guardian able to provide informed consent

Exclusion Criteria:

* Any acute or chronic condition that, in the investigator's opinion, significantly interferes with assessments and/or motor development.
* Participation in a therapeutic trial.
* Lack of internet connection.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Digital Mobility Monitoring Compliance | 4 weeks of recording periods every 3 months over 2 years
  Measure of participant adherence to wearing the Syde® device: total recording time.
Digital Mobility Monitoring Compliance | 4 weeks of recording periods every 3 months over 2 years
  Measure of participant adherence to wearing the Syde® device: number of valid recording days (≥4 hours)
Digital Mobility Monitoring Compliance | 4 weeks of recording periods every 3 months over 2 years
  Measure of participant adherence to wearing the Syde® device: time to reach 50 and 180 hours of recording.
Digital Mobility Monitoring Compliance | 1 day of recording periods every month over 2 years
  Measure of participant adherence to wearing the MAIJU® device using total recording time.
Walking Pattern Characteristics | 4 weeks of recording periods every 3 months over 2 years
  Analysis of walking sequences: maximal walking sequence duration
Walking Pattern Characteristics | 4 weeks of recording periods every 3 months over 2 years
  Analysis of walking sequences: maximal distance walked in a single sequence.
Walking Pattern Characteristics | 4 weeks of recording periods every 3 months over 2 years
  Analysis of walking sequences: maximal 30-minute walking distance.
Reliability | Baseline, 1 year, 2 years.
  Inter Class Correlation (ICC2K) when comparing the first and the second half of recordings that includes more than 100 hours AND more than 2000 steps
Group Differences in Digital Variables | Age 2, 3 and 4 years
  Comparison of digital mobility metrics across subgroups defined by the number of SMN2 copies (SMA patients) and age's symptom appearance with
  1. Patients with SMA symptoms at treatment initiation
  2. Patients with 2 copies of SMN2 and no symptoms at treatment initiation
  3. Patients with 3 copies of SMN2 and no symptoms at treatment initiation
  4. Patients with 4 copies of SMN2
  5. Healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Dangouloff, PhD, Principal Investigator — University of Liege; Laurent Servais, MD, PhD, Study Director — University of Liege
Locations (1):
- Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No